CLINICAL TRIAL: NCT01706692
Title: Long-Term Benefits and Safety of Systemic Psoriasis Therapy: Swiss Registry on the Treatment of Psoriasis With Biologics and Systemic Therapeutics
Brief Title: Swiss Dermatology Network of Targeted Therapies (SDNTT)
Acronym: SDNTT
Status: Recruiting | Type: Observational
Sponsor: Swiss Dermatology Network for Targeted Therapies (Other)
Responsible Party: Sponsor
Other Study IDs: IMM 10-0138; P21007224R; CNTO1275PSO4028; AG110401-IIR (Other Grant/Funding Number: AbbVie, Almirall, Janssen Pharmaceutica, Eli Lilly, UCB)
Record Dates: First submitted 2012-09-19; First posted 2012-10-15 (Estimated); Last update posted 2024-11-29 (Actual); Status verified 2024-11

CONDITIONS: Psoriasis
Keywords: Methotrexate; Acitretin; Cyclosporine A; Systemic PUVA; Infliximab; Adalimumab; Etanercept; Ustekinumab; Fumaric acids; Psoriasis; Psoriatic arthritis; Skin disease
MeSH Terms: conditions — Psoriasis; Arthritis, Psoriatic; Skin Diseases | interventions — Adalimumab; Etanercept; Infliximab; Ustekinumab; Cyclosporine; Methotrexate

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (8):
- Adalimumab: Intervention: Biological: Adalimumab, all dosages, frequencies and durations prescribed
  Interventions: Biological: Adalimumab
- Etanercept: Intervention: Biological: Etanercept, all dosages, frequencies and durations prescribed
  Interventions: Biological: Etanercept
- Infliximab: Intervention: Biological: Infliximab, all dosages, frequencies and durations prescribed
  Interventions: Biological: Infliximab
- Ustekinumab: Intervention: Biological: Ustekinumab, all dosages, frequencies and durations prescribed
  Interventions: Biological: Ustekinumab
- Cyclosporine A: Intervention: Drug: conventional systemic: Cyclosporine A, all dosages, frequencies and durations prescribed
  Interventions: Drug: Cyclosporine A
- Fumaric acids: Intervention: Drug: conventional systemic: Fumaric acids, all dosages, frequencies and durations prescribed
  Interventions: Drug: Fumaric acids
- Methotrexate: Intervention: Drug: conventional systemic: Methotrexate, all dosages, frequencies and durations prescribed
  Interventions: Drug: Methotrexate
- Other anti-psoriatic systemic treatments: e.g.: Intervention: Drug: conventional systemic: Acitretin or Systemic phototherapy (PUVA), all dosages, frequencies and durations prescribed
  Interventions: Drug: Other anti-psoriatic systemic treatments

INTERVENTIONS:
Biological: Adalimumab — all dosages, frequencies and durations prescribed
  Other Names: Humira
  Groups: Adalimumab
Biological: Etanercept — all dosages, frequencies and durations prescribed
  Other Names: Enbrel
  Groups: Etanercept
Biological: Infliximab — all dosages, frequencies and durations prescribed
  Other Names: Remicade
  Groups: Infliximab
Biological: Ustekinumab — all dosages, frequencies and durations prescribed
  Other Names: Stelara
  Groups: Ustekinumab
Drug: Cyclosporine A — all dosages, frequencies and durations prescribed
  Groups: Cyclosporine A
Drug: Fumaric acids — all dosages, frequencies and durations prescribed
  Groups: Fumaric acids
Drug: Methotrexate — all dosages, frequencies and durations prescribed
  Groups: Methotrexate
Drug: Other anti-psoriatic systemic treatments — all dosages, frequencies and durations prescribed
  Groups: Other anti-psoriatic systemic treatments

SUMMARY:
The purpose of this study is to evaluate the long-term course of patients with psoriasis and psoriatic-arthritis in systemic treatments such as, methotrexate, cyclosporin A, fumaric acids, acitretin, systemic PUVA, etanercept, infliximab, adalimumab and ustekinumab. A patient will be included at first initiation of the treatment and will remain in the registry for 10 years, regardless of subsequent therapy.

The registry will also evaluate safety clinical outcomes and health related quality of life.

DETAILED DESCRIPTION:
Treatment of moderate to severe Psoriasis (Pso) and Psoriasis-Arthritis (PsA) in Switzerland is largely performed with systemic therapies. This includes conventional systemic therapy such as fumaric acids, methotrexate, cyclosporin A, retinoids, systemic PUVA, Acitretin and biological treatments such as etanercept, infliximab, adalimumab and within a pre-registration program ustekinumab. While short- and middle-term efficacy of most systemic treatments has been shown in clinical studies (and is incorporated in international guidelines), knowledge about long-term outcomes, optimal treatment and effectiveness under real-world conditions is still missing. SDNTT, the Swiss registry on the treatment of moderate to severe Pso and PsA documents the long-term course of patients being administered a defined biologic or conventional systemic drug. Following outcomes are observed: Effectiveness on the long-term, of combined/alternating treatments and under comorbidity conditions; patient-defined benefits and quality of life, maintenance dosages, prediction of response and safety.

The study evaluates the long-term course of patients with Pso and PsA in systemic treatments. A patient will be included at first initiation of the treatment and will remain in the registry for 5 years, regardless of subsequent therapy. Nationwide, initially 35 (long-term approx. 50-80) dermatologic practices and hospital ambulances with expertise in systemic and biologic treatment will consecutively enroll patients. Follow-ups will be every 3 months, comprising patient and treatment characteristics, clinical parameters, patient-defined benefit, quality of life and adverse events. Standardized questionnaires will be addressed to the patient and to the dermatologist 12 times at the dermatologic centres. In interim intervals, patients are directly contacted another 9 times by mail.

ELIGIBILITY:
Inclusion Criteria:

* Patients with diagnosis of plaque-type psoriasis or psoriasis arthritis confirmed by a dermatologist,
* age ≥ 18,
* Being administered a specific biologic/conventional systemic drug for the first time
* Sufficient language skills (German, French, Italian and English) for the informed consent to participate
* Informed consent to participate

Exclusion Criteria:

* Lack of informed consent
* Patients being participants of clinical trials at the day of registration to the registry (if a patient is included into a clinical trial during the registry follow-ups, the patient data will be recorded, but analyzed separately)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Any patient with psoriasis or psoriatic-arthritis meeting the inclusion criteria and not meeting the exclusion criteria will be eligible to participate in this registry.
Sampling Method: Non-Probability Sample
Enrollment: 1121 (Estimated)
Dates: Start 2011-02; Primary Completion 2032-03-15 (Estimated); Study Completion 2032-03-15 (Estimated)

PRIMARY OUTCOMES:
Psoriasis Area Severity Index (PASI) | every 6 months for 10 years
  To evaluate clinical outcome of patients exposed to conventional systemic or biologic therapy for psoriasis/psoriatic-arthritis

SECONDARY OUTCOMES:
Dermatology Life Quality Index (DLQI) | every 6 months for 10 years
  To evaluate health related quality of life of patients exposed to conventional systemic or biologic therapy for psoriasis/psoriatic-arthritis

OTHER OUTCOMES:
Adverse and serious adverse events | 10 years
  Risk for adverse events and serious adverse events for patients exposed to conventional systemic or biologic therapy for psoriasis/psoriatic-arthritis

CONTACTS AND LOCATIONS:
Overall Officials: Alexander Navarini, Prof Dr med, Principal Investigator — Swiss Society of Dermatology and Venereology (SSDV); Julia-Tatjana Maul, PD Dr med, Principal Investigator — Swiss Society of Dermatology and Venereology (SSDV)
Locations (6):
- Switzerland (6):
  - Aarau Cantonal Hospital, Aarau
  - Basel University Hospital, Basel
  - Inselspital - Bern University Hospital, Bern
  - Centre Hospitalier Universitaire Vaudois (CHUV), Lausanne
  - St. Gallen Cantonal Hospital, Sankt Gallen
  - Zurich University Hospital, Zurich

REFERENCES:
- See also: SDNTT — https://www.sdntt.ch
- See also: German registry PsoBest — http://www.psobest.de/